CLINICAL TRIAL: NCT06221644
Title: Synapse Alterations in MSA Patients
Status: Completed | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: 20240113
Record Dates: First submitted 2024-01-15; First posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Multiple System Atrophy
Keywords: synaptic density; PET; SV2A
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MSA patients group: The patient cohort consisted of 30 MSA-C and 30 MSA-P cases, diagnosed according to the 2008 Second Consensus Criteria and confirmed by two experienced neurologists
  Interventions: Diagnostic Test: [18F]SynVesT-1 PET/CT
- healthy controls (HCs) group: 30 gender and age-matched HCs were included
  Interventions: Diagnostic Test: [18F]SynVesT-1 PET/CT

INTERVENTIONS:
Diagnostic Test: [18F]SynVesT-1 PET/CT — 60 MSA patients (30 MSA-P subtype and 30 MSA-C subtype) and 30 age-matched healthy controls (HCs) underwent [18F]SynVesT-1 PET/CT for synaptic density assessment

SUMMARY:
Synaptic loss has been implicated in various neurodegenerative conditions, yet its understanding in multiple system atrophy (MSA) remains limited.

The aim of this study was to examine spatial synaptic density alterations in MSA patients and evaluate the potential of [18F]SynVesT-1 PET as an imaging biomarker for MSA in both diagnosis and monitoring disease severity.

DETAILED DESCRIPTION:
60 MSA patients (30 MSA-P subtype and 30 MSA-C subtype) and 30 age-matched healthy controls (HCs) underwent [18F]SynVesT-1 PET/CT for synaptic density assessment. Visual, voxel, and volumetric region-of-interest (VOI) analyses were employed to elucidate synaptic density patterns in the MSA brain and establish visual diagnostic criteria. VOI-based computer-assisted analyses were utilized to develop diagnostic models for MSA.

ELIGIBILITY:
Inclusion Criteria:

The MSA patient were diagnosed according to the 2008 Second Consensus Criteria and confirmed by two experienced neurologists.

Exclusion Criteria:

encompassed MRI contraindications, a history of epilepsy, stroke, or brain surgery, intracranial organic lesions unrelated to MSA, usage of levetiracetam or brivaracetam, and a history of alcohol or drug abuse

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 60 patients diagnosed with MSA were recruited. The patient cohort consisted of 30 MSA-C and 30 MSA-P cases, diagnosed according to the 2008 Second Consensus Criteria and confirmed by two experienced neurologists. Additionally, 30 gender and age-matched HCs were included.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Spatial synaptic density alterations in MSA patients | 10 months
  To examine spatial synaptic density alterations in MSA patients
[18F]SynVesT-1 PET as an imaging biomarker for MSA | 10 months
  evaluate the potential of [18F]SynVesT-1 PET as an imaging biomarker for MSA

CONTACTS AND LOCATIONS:
Overall Officials: Shuo Hu, Study Chair — Shuo Hu
Locations (1):
- Jian Li, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No